CLINICAL TRIAL: NCT02607943
Title: Insulin Glargine Versus Regular Insulin Based Regimens in Glycemic Control After Acute Stroke: A Multi-center, Randomized Control Study
Brief Title: Insulin Glargine Versus Regular Insulin Based Regimens in Glycemic Control After Acute Stroke
Acronym: ICAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201504075MINC
Record Dates: First submitted 2015-11-04; First posted 2015-11-18 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Acute Stroke; Hyperglycemia
Keywords: acute stroke; hyperglycemia; regular insulin; long-acting insulin
MeSH Terms: conditions — Stroke; Hyperglycemia; Insulin Resistance | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Glargine (Experimental): subcutaneous long acting basal insulin (insulin glargine) with added short acting regular insulin to correct hyperglycemic events
  Interventions: Drug: Insulin Glargine
- Regular Insulin (Active Comparator): short acting regular insulin pre-meal with added NPH at bed time if start eating
  Interventions: Drug: Regular Insulin

INTERVENTIONS:
Drug: Insulin Glargine — Insulin Glargine Versus Regular Insulin Based Regimens in Glycemic Control
  Other Names: Lantus
  Arms: Insulin Glargine
Drug: Regular Insulin — Insulin Glargine Versus Regular Insulin Based Regimens in Glycemic Control
  Arms: Regular Insulin

SUMMARY:
Hyperglycemia is common during acute ischemic stroke. However, the optimal strategy to control hyperglycemia during acute ischemic stroke has not been established. The object of this multicenter randomized controlled study is to determine the efficacy and safety of early initiation of subcutaneous once-daily insulin glargine, in comparison with regular insulin, based on a protocolized sliding scale regimen to achieve proper sugar control in acute stroke patients with hyperglycemia admitted to the intensive care unit.

DETAILED DESCRIPTION:
Study Rationale: Hyperglycemia is common during acute ischemic stroke. It has been shown that persistent in-hospital hyperglycemia during the first 24 hours (h) after stroke is associated with worse outcomes than normoglycemia. However, the optimal strategy to control hyperglycemia during acute ischemic stroke has not been established.

Aims: The object of this multicenter randomized controlled study is to determine the efficacy and safety of early initiation of subcutaneous once-daily insulin glargine, in comparison with regular insulin, based on a protocolized sliding scale regimen to achieve proper sugar control in acute stroke patients with hyperglycemia admitted to the intensive care unit (ICU).

Design: This is a 3-year, randomized, multicenter trial. Approximate 120 hyperglycemic acute stroke patients will receive either (a) subcutaneous long acting basal insulin (insulin glargine) with added short acting regular insulin to correct hyperglycemic events or (b) short acting regular insulin pre-meal with added NPH at bed time if start eating, for 72 h, starting within 24 h of stroke symptom onset. The inclusion criteria are patients who admitted to stroke ICU within 24 hours of acute stroke onset and have repeated random blood glucose >200 mg/dL with a 2 hours interval. The exclusion criteria include patients with age <20 years, pregnancy, shock, severe infection, end stage renal disease requiring dialysis, type I DM or current steroid usage. Capillary blood glucose will be measured every 4-hours to adjust the next insulin dose. Glucometric parameters will also be analyzed by continuous blood glucose monitoring system. 10 ml blood and same amount of urine from 24 hours urine collection will be collected every day for further measurement of a variety of blood inflammatory markers and urine catecholamine levels.

Study outcomes: The primary endpoint is the percentage of time in the range of 80-180 mg/dL during the sugar monitoring period. The secondary endpoints include: (1) good functional outcome at 3 months post stroke (modified Rankin Scale <2), (2) stroke in evolution, (3) 24 hours blood glucose variability via continuous glucose monitoring, and (4) blood and urine biomarkers.

In summary, this trial will provide important novel information about preferred management of acute ischemic stroke patients with hyperglycemia. It will determine the potential benefits and risks of application of long acting basal insulin during very early stage of acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to stroke ICU within 24 hours of acute stroke onset and have repeated random blood glucose >200 mg/dL with a 2 hours interval

Exclusion Criteria:

* Patients with age <20 years,
* pregnancy,
* shock, severe infection, end stage renal disease requiring dialysis,
* type I DM or current steroid usage.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of time in the range of 80-180 mg/dL during the sugar monitoring period | 72 hours after recruitment

SECONDARY OUTCOMES:
Good functional outcome at 3 months post stroke | 3 months after stroke
  Good functional outcome is defined as modified Rankin Scale <2
Stroke in evolution | one week after stroke onset
  Stroke in evolution is defined as an increase in the National Institutes of Health Stroke Scale (NIHSS) score of ≥ 2 points excluding other attributable medical or systemic causes.
Blood glucose variability via continuous glucose monitoring | 72 hours after recruitment
  Blood glucose is monitored 24 hours per day via continuous glucose monitoring for 72 hours after recruitment to evaluate the variability.
Blood biomarkers | 72 hours after recruitment
  Blood biomarkers include soluble form of receptor for glycation end-product (sRAGE), high mobility group box 1(HMGB1), heat shock protein 70 (HSP 70), C-reactive protein (CRP), D-dimer, fibrinogen
Urine biomarkers | 72 hours after recruitment
  Urine biomarkers include catecholamines such as normetanephrine and vanillylmandelic acid (VMA)

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Shing Jeng, MD. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tang SC, Shih SR, Lin SY, Chen CH, Yeh SJ, Tsai LK, Yang WS, Jeng JS. A randomized trial to investigate the efficacy and safety of insulin glargine in hyperglycemic acute stroke patients receiving intensive care. Sci Rep. 2021 Jun 1;11(1):11523. doi: 10.1038/s41598-021-91036-2. PMID 34075142